CLINICAL TRIAL: NCT02848014
Title: The Effects of Interventions Aiming at Optimizing Expectations and Inducing Positive Emotions After an Acute Stressor on Subjective and Objective Stress Paramaters
Brief Title: The Effects of Interventions Aiming at Optimizing Expectations and Inducing Positive Emotions After an Acute Stressor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-08k
Record Dates: First submitted 2016-06-29; First posted 2016-07-28 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Expectation (Experimental): Participants are asked to think and write about ways how they can positively influence/control the stress during stress induction. They also can think of strategies they used in their past. The purpose of this arm is to improve participants' personal control expectations.
  Interventions: Behavioral: Writing task
- Emotion (Experimental): Participants in this group are asked to write a gratitude-letter to a person they want to thank. The purpose of this arm is to foster positive emotions.
  Interventions: Behavioral: Writing task
- Control (Active Comparator): Participants in this group are asked to do a neutral writing task. The task is to write a protocol of yesterday's to-dos.
  Interventions: Behavioral: Writing task

INTERVENTIONS:
Behavioral: Writing task

SUMMARY:
The purpose of the study is to determine whether a short psychological intervention aiming at optimizing expectations is able to foster positive emotions and whether an intervention inducing positive emotions is able improve participants' expectations. Furthermore, the investigators will examine whether both interventions are effective in buffering the stress response after an acute stressor in a healthy sample compared to a control condition.

ELIGIBILITY:
Inclusion Criteria:

* fluent in German language

Exclusion Criteria:

* chronic disease
* mental disease
* the evening before the day of the experiment until end of the experiment (the next day): caffeine, alcohol, intensive physical exercise, chewing gum
* acute hay fever
* current intake of psychotropic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change in personal control expectation (Item of the Brief IPQ) | Pre-intervention (baseline; T0) vs. Post-intervention (25 minutes after baseline assessment; T1)

SECONDARY OUTCOMES:
Change in emotions (PANAS) | Pre-intervention (baseline; T0) vs. Post-intervention (25 minutes after baseline assessment; T1)
Subjective stress ratings | directly after completing the stress induction (approximately 50 minutes after baseline assessment; T2)
  Questionnaire items
Change in Cortisol levels (saliva sample) | Pre-intervention (baseline; T0) vs.Post-intervention (25 minutes after baseline assessment; T1), directly (T2), 15 min (T3) and 30 min (T4) after stress induction
  directly (T2), 15 min (T3) and 30 min (T4) after stress induction = 50 min, 65 min and 80 min after baseline assessment
Change in Alpha-Amylase levels (saliva sample) | Pre-intervention (baseline; T0) vs. Post-intervention (25 minutes after baseline assessment; T1), directly (T2), 15 min (T3) and 30 min (T4) after stress induction
  directly (T2), 15 min (T3) and 30 min (T4) after stress induction = 50 min, 65 min and 80 min after baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Professor, Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany